CLINICAL TRIAL: NCT00246181
Title: Phase I and II Study Of Stereotactic Body Radiotherapy in Medically Unresectable Patients With Stage 1 NSCLC
Acronym: SBF-NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jill Deluca (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Jill Deluca, Research Coordinator, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9910-35
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung cancer; stereotactic body radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: radiation therapy — Patients will receive 3 fractions

SUMMARY:
This clinical trial involves a radiation treatment called stereotactic radiotherapy in non-small cell lung cancer patients who have been determined to be ineligible for surgery. This treatment differs from conventional radiotherapy in the number of treatments, the radiation dose given per treatment, and the way the radiation beams are directed toward the cancer.

DETAILED DESCRIPTION:
The most common treatment for early stage lung cancers is to remove the cancer with surgery. Patients with serious underlying health problems like emphysema, diabetes, or heart disease who develop an early stage lung cancer may not be eligible for the standard surgical treatment. The most common alternative to surgery is conventional radiation treatment called fractionated radiotherapy. "Fractionated radiotherapy" means several weeks of treatment with daily radiation sessions. While this treatment is sometimes successful at killing the cancer, it is not as effective as surgery and may significantly damage the surrounding lung tissue.

Newer treatments using radiotherapy have been developed and used for patients with metastases (spreading cancer) to the lungs. Stereotactic radiotherapy uses a frame to guide highly focused beams of radiation at the cancer while avoiding the normal surrounding tissue. Stereotactic radiotherapy also uses a higher daily dose of radiation. The higher daily dose may be more effective than conventional radiotherapy at killing cancer cells and may also decrease side effects.

ELIGIBILITY:
Inclusion Criteria:

Consistent with most therapeutic oncology trials, patients are not actively "recruited," but are screened by their physician for appropriate clinical trial(s) at the time of their routine clinic visit.

All patients must be willing and capable to provide informed consent to participate in the protocol.

Eligible patients must have appropriate staging studies identifying them as AJCC stage I (T1 or T2, N0, M0) primary lung carcinoma. The patient should not have direct evidence of regional or distant metastases after appropriate staging studies. Histologic confirmation will be required by either biopsy or cytology. The following primary cancer types are eligible: Squamous cell carcinoma, Adenocarcinoma, Large cell carcinoma, bronchioloalveolar cell carcinoma or non-small cell; not otherwise specified.

The primary tumor must be deemed technically resectable by an experienced thoracic cancer clinician, with a reasonable possibility of obtaining a gross total resection with negative margins (defined as a potentially curative resection, PCR); however, the patient should have underlying physiological medical problems that would prohibit a PCR due to a low probability of tolerating general anesthesia, the operation, the post-operative recovery period, or the removal of adjacent functioning lung. Standard "cut-off " guidelines regarding surgical resection of NSCLC include the following: Baseline FEV1 <40%, post-operative predicted FEV1 <30%, severely reduced diffusion capacity, baseline hypoxemia and/or hypercapnia and exercise oxygen consumption <50% predicted.

Patients who refuse a PCR due to preference, ideology, emotional or psychological issues, mental illness, or inability to give consent for the PCR and who have no specific accepted medical contraindications for the PCR are not eligible.

Eligible patients should not have had previous lung or mediastinal radiotherapy.

There must be no plans for the patient to receive other concomitant antineoplastic therapy while on this protocol. Patients who have received chemotherapy within 8 weeks of the start date of study are ineligible.

Patients must be able to fit inside the stereotactic body frame and able to undergo a CT or MRI scan in the frame.

The patient's primary tumor must not be larger than 7.0 cm in greatest dimension.

Patients with active systemic, pulmonary, or pericardial infection are ineligible.

Pregnant or lactating women are ineligible. Women/men of reproductive potential may not participate unless they agreed to use an effective contraceptive method such as condom/diaphragm and spermicidal foam, intrauterine device (IUD), or prescription birth control pills.

Patients must be past their 18th birthday at time of registration. Karnofsky performance status > 60.

-

Exclusion Criteria:

See inclusion criteria.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 1999-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The purposes of this research study are (1) to find the highest dose of stereotactic radiotherapy that can safely be used for treatment of early stage non-small cell lung cancer. | 5 years from enrollment completion

SECONDARY OUTCOMES:
(2) to see what effects (good and bad) stereotactic radiotherapy has on patients and their cancer. | 5 years from completion enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Ronald McGarry, MD, Principal Investigator — Indiana University - Department of Radiation Oncology; Achilles Fakiris, MD, Principal Investigator — Indianan University
Locations (1):
- Indiana University, Department of Radiation Oncology, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Henderson M, McGarry R, Yiannoutsos C, Fakiris A, Hoopes D, Williams M, Timmerman R. Baseline pulmonary function as a predictor for survival and decline in pulmonary function over time in patients undergoing stereotactic body radiotherapy for the treatment of stage I non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2008 Oct 1;72(2):404-9. doi: 10.1016/j.ijrobp.2007.12.051. Epub 2008 Apr 18. PMID 18394819
- See also: Link to Department of Radiation Oncology — http://www.medicine.iu.edu/body.cfm?id=4491